CLINICAL TRIAL: NCT05628454
Title: Comparison of Three Different Puncture Techniques in EBUS-TBNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: BFH20221019005
Record Dates: First submitted 2022-11-06; First posted 2022-11-28 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer; Sarcoidosis; Tuberculosis
MeSH Terms: conditions — Lung Neoplasms; Sarcoidosis; Tuberculosis | interventions — Suction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The operator knows which puncture technique to be used, but the subject and the outcomes assessor does not know the technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EBUS-TBNSP (Experimental): The slow-pull capillary technique was performed as follows: after identification and measurement of the target lymph node, a needle was used to puncture the lymph node with the stylet in place.At the same time, the stylet was slowly and continuously pulled to create weak negative pressure.
  Interventions: Procedure: Endobronchial ultrasound-guided transbronchial needle Slow-pull capillary sampling
- EBUS-TBNA (Experimental): The operation steps are the same as above, but the negative pressure device of 10ml syringe is connected behind the puncture needle.
  Interventions: Procedure: Endobronchial ultrasound-guided transbronchial needle aspiration
- EBUS-TBNCS (Experimental): The operation steps are the same as above, but there is no negative pressure device behind the puncture needle
  Interventions: Procedure: Endobronchial ultrasound-guided transbronchial needle capillary sampling

INTERVENTIONS:
Procedure: Endobronchial ultrasound-guided transbronchial needle Slow-pull capillary sampling — The slow-pull capillary technique was performed as follows: after identification and measurement of the target lymph node, a needle was used to puncture the lymph node with the stylet in place.At the same time, the stylet was slowly and continuously pulled to create weak negative pressure.
  Other Names: Slow-pull capillary technique
  Arms: EBUS-TBNSP
Procedure: Endobronchial ultrasound-guided transbronchial needle aspiration — The operation steps are the same as above, but the negative pressure device of 10ml syringe is connected behind the puncture needle.
  Other Names: Standard suction
  Arms: EBUS-TBNA
Procedure: Endobronchial ultrasound-guided transbronchial needle capillary sampling — The operation steps are the same as above, but there is no negative pressure device behind the puncture needle
  Other Names: Fine needle sampling without suction
  Arms: EBUS-TBNCS

SUMMARY:
The purpose of this study was to compare the accuracy and sensitivity of slow-pull capillary technique, traditional suction aspiration and non negative pressure puncture in the diagnosis of mediastinal and/or hilar lymph node enlargement by ultrasound bronchoscopic lymph node biopsy.

DETAILED DESCRIPTION:
EBUS-TBNA has been widely used in the diagnosis of diseases involving lung hilar and mediastinal lymph node enlargement.But different puncture methods are still controversial. Research shows that there was no significant difference in sample adequacy, diagnostic specificity and accuracy between the no negative pressure aspiration and traditional negative pressure aspiration technique.Slow-pull capillary technique is a relatively new operating method of endoscopic ultrasound guided fine needle biopsy in recent years. At present, this technology is widely used in pancreatic space occupying lesions. Compared with the traditional negative pressure aspiration method, our previous retrospective study found that the slow-pull capillary technique can improve the diagnostic accuracy of patients. Therefore, the purpose of this study is to prospectively and randomly compare the advantages and disadvantages of three puncture methods in EBUS-TBNA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80years
* Chest computed tomography showing hilar or mediastinal lymph node enlargement
* No contraindications for bronchoscopy
* Signed informed consent provided by the patient
* Disease needs to be diagnosed through the EBUS-TBNA

Exclusion Criteria:

* Severe coagulation dysfunction
* Severe cardiopulmonary dysfunction
* Acute asthma attack or massive haemoptysis
* Poor general condition
* Physical weakness without tolerance for anaesthesia or allergy to narcotic drug
* Disease can be diagnosed by other less invasive methods (such as skin or peripheral superficial lymph node biopsy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of three different puncture methods according to pathological diagnosis | 6 months
  The final pathological diagnosis was based on all available cytological and histological samples. In cases with negative pathological results , we continue to follow up the patients for ⩾6months.

SECONDARY OUTCOMES:
Blood contamination of samples | 1 week
  Blood contamination was categorized as follows: low (no or few blood cells influencing the diagnosis), moderate (sample partially obscured by blood cells, but pathological diagnosis possible), and high (large numbers of blood cells, rendering pathological diagnosis difficult)
Bleeding of operation | 1 week
  There are three levels of bleeding:Small amount of bleeding（Ⅰ）: Bleeding can stop spontaneously without continuous suction.Moderate bleeding（Ⅱ）: Continuous suction is required, and epinephrine or ice salt water is used locally to stop bleeding.Massive bleeding（Ⅲ）: Patients who need to be used balloon compression, interventional treatment, or blood transfusion treatment or even died of asphyxia due to bleeding.
Acquisition of tissue core of three different puncture methods according to the judgment of the pathologist | 1 week
  Tissue cores were immersed in formalin solution and subjected to histopathological examination. In the absence of a tissue core, the contents were pressed onto a glass slide, immersed in 96% methanol for ⩾10min and subjected to cytopathological examination.Some methods may only obtain cytological specimens, while others may obtain tissue cores. Tissue cores are better for pathologists to diagnose.

CONTACTS AND LOCATIONS:
Overall Officials: Yanjun Wu, Principal Investigator — Beijing Friendship Hospital; Zhigang Yao, Study Director — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wu Y, Xu R, Duan X, Deng Y, Yu G, He X, Yao Z. Comparison of three different puncture techniques for endobronchial ultrasound transbronchial needle aspiration: a single-center, prospective, randomized controlled study. BMC Pulm Med. 2025 Sep 30;25(1):437. doi: 10.1186/s12890-025-03917-1. PMID 41029266